CLINICAL TRIAL: NCT04384133
Title: The Prevalence of Small Airways Dysfunction In COPD Patients and The Impact on COPD Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sibel Naycı (Other)
Collaborators: Mersin University (Other)
Responsible Party: Sponsor-Investigator, Sibel Naycı, Clinical Professor of Pulmonology, Mersin University
Organization: Mersin University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-2-TP3-3539-2
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COPD; Small Airway Disease
Keywords: COPD; Small Airway Dysfunction; Impulse oscillometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fractional Exhaled Nitric Oxide Testing; Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COPD group (Other): Impulse oscillometric pulmonary function tests and spirometric pulmonary function test will be performed.To evaluate the degree of disease inflammation and phenotype, nitric oxide measurements will be made in the breath air with fractional exhaled nitric oxide (FENO) device. Blood eosinophil values will be examined. Thorax computed tomography will be performed to evaluate small airway dysfunction. To assess symptom control in patients with COPD, a dyspnea scale of mMRC will be administered. The COPD assessment test (CAT) will be applied to measure the quality of life. All participants will be followed for 1 year to record the number of exacerbations requiring emergency and hospital admissions for COPD.
  Interventions: Diagnostic Test: Impulse oscillometry; Diagnostic Test: Spirometric pulmonary function test; Diagnostic Test: Fractional exhaled nitric oxide (FENO) test; Diagnostic Test: Thorax Computed Tomography; Diagnostic Test: Blood eosinophil level; Other: CAT; Other: mMRC
- Healthy control group with a history of smoking (Other): Impulse oscillometric pulmonary function test, spirometric pulmonary function test and chest x ray will be performed.
  Interventions: Diagnostic Test: Impulse oscillometry; Diagnostic Test: Spirometric pulmonary function test; Diagnostic Test: Chest X Ray
- Healthy control group with no smoking history (Other): Impulse oscillometric pulmonary function test, spirometric pulmonary function test and chest x ray will be performed.
  Interventions: Diagnostic Test: Impulse oscillometry; Diagnostic Test: Spirometric pulmonary function test; Diagnostic Test: Chest X Ray

INTERVENTIONS:
Diagnostic Test: Impulse oscillometry — Impulse oscillometry is a pulmonary function test. During the test, the participant is told to breathe normally.
Diagnostic Test: Spirometric pulmonary function test — In the spirometric pulmonary function test, the participant is asked to perform respiratory maneuvers such as breathing deeply.
Diagnostic Test: Fractional exhaled nitric oxide (FENO) test — In the FENO test, the participant is asked to perform respiratory maneuvers such as breathing deeply.
  Arms: COPD group
Diagnostic Test: Thorax Computed Tomography — Computed tomography is a radiological examination.
  Arms: COPD group
Diagnostic Test: Chest X Ray — Chest X ray is a radiological examination.
  Arms: Healthy control group with a history of smoking; Healthy control group with no smoking history
Diagnostic Test: Blood eosinophil level — A tube of blood will be drawn from the participant.
  Arms: COPD group
Other: CAT — It consists of 8 questions.
  Arms: COPD group
Other: mMRC — It is the scale used to measure the severity of shortness of breath.
  Arms: COPD group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a worldwide prevalent disease. During recent years, increasing attention has been directed to the importance of the contribution of small airways in respiratory diseases. The small airways (usually defined as those with an internal diameter of <2 mm) are recognized as the major site of resistance to airflow in obstructive lung disease. Although small airway disease is known in chronic airway diseases, the importance of small airway dysfunction on disease control, exacerbations and quality of life, and the importance of taking place among treatable targets is not clear. Therefore, our aim in the study is to determine the frequency of small airway dysfunction in COPD. Our secondary aim is to evaluate the role of small airway dysfunction in disease severity, disease phenotypes, disease control, quality of life and its effect on predicting the risk of exacerbation and its role among treatable targets in chronic airway diseases.

DETAILED DESCRIPTION:
This is a prospective cross-sectional interventional design. 100 COPD patients who applied to Mersin University Faculty of Medicine Hospital Chest Diseases Clinic between 01.10.2019-01.04.2020 will be taken. 35 healthy participants with smoking history and 35 healthy participants without smoking history who were admitted to our clinic within the same date range will be taken as control group. Impulse oscillometric pulmonary function tests will be performed to all participants. Thorax computed tomography will be performed to evaluate small airway dysfunction. To evaluate the degree of disease inflammation and phenotype in COPD patients, nitric oxide measurements will be made in the breath air with fractional exhaled nitric oxide (FENO) device. The blood eosinophil level will be studied to determine the COPD phenotype. To assess symptom control in patients with COPD, mMRC(Modified Medical Research Council) dyspnea scale will be administered. The COPD assessment test (CAT) will be applied to measure the quality of life. All patients will be followed for 1 year to record the number of exacerbations requiring emergency and hospital admissions for COPD. The effect of small airway dysfunction on the disease severity and control degree, disease phenotypes and quality of life, and the effect on the risk of exacerbation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

COPD group

* Participants who applied to the chest diseases clinic of Mersin University Hospital, between October 1, 2019 and April 1, 2020
* Participants who were diagnosed COPD with spirometry test
* Reading and signing Informed Consent Form
* Participants must be older than 18 years

Healthy control group with a history of smoking

* To apply to the chest diseases clinic of Mersin University Hospital between October 1, 2019 and April 1, 2020
* Reading and signing informed consent form
* Participants must be older than 18 years
* Must have no lung disease
* Must have 10 packs / year or more than 10 packs / year smoking history

Healthy control group without smoking history

* To apply to the chest diseases clinic of Mersin University Hospital between October 1, 2019 and April 1, 2020
* Reading and signing informed consent form
* Participants must be older than 18 years
* Must have no lung disease
* Must have no smoking history

Exclusion Criteria:

* Participants who do not sign the Informed Consent Form
* Under the age of 18 years
* Pregnant women
* Participants who with a history of cancer in the past 5 years
* Participants who previously had lung surgery
* Participants who with Interstitial Lung Disease
* Participants who with respiratory muscle disease
* Participants who with active pulmonary tuberculosis
* Participants who can not perform respiratory function tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Small airway dysfunction will be evaluated by performing impulse oscillometry test. | through study completion, an average of 1 year
  Respiratory resistance at 5 and 20 Hz (R5 and R20, respectively) will be used for the analyses. R5 and R20 are regarded as reflecting total and proximal airway resistance, respectively, and the fall in resistance from R5 to R20 (R5-R20) will used as a surrogate for the resistance of small airways.
Small airway dysfunction will be evaluated by thorax computed tomography. | through study completion, an average of 1 year
  Indirect changes caused by the small airways on the lung parenchyma will be detected by computed tomography (CT).
Small airway dysfunction will be evaluated by body plethysmography test. | through study completion, an average of 1 year
  Residual volume (RV) and total lung capacity (TLC) will be measured by body plethysmography test to determine small airway dysfunction.
Symptoms will be evaluated by Modified Medical Research Council Dyspnea Scale (mMRC). | through study completion, an average of 1 year
  The mMRC (Modified Medical Research Council) scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing.
The number of moderate and severe exacerbations over a 1 year period will be recorded. | through study completion, an average of 1 year
  In the COPD group, each participant will be followed for 1 year in terms of recording exacerbations.
Forced expiratory volume in 1 second (fev1) change will be evaluated by spirometric pulmonary function test. | through study completion, an average of 1 year
  Forced expiratory volume in 1 second (fev1) change over one year period will be evaluated with spirometric pulmonary function test during recruitment and 1st year of follow-up.

SECONDARY OUTCOMES:
Fractional Exhaled Nitric Oxide (FENO) test will be used as an indicator of inflammation. | through study completion, an average of 1 year
  FENO test is indirect measurements of inflammation, as used in clinical practice.
Complete blood count ( CBC) test will be used as an indicator of inflammation. | through study completion, an average of 1 year
  Blood eosinophil levels will be recorded.
Quality of life will be evaluated by COPD Assessment Test (CAT). | through study completion, an average of 1 year
  COPD Assessment Test (CAT) contains 8 questions. In each question, the minimum value is zero and the maximum value is five points. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Nayci, Prof.Dr., Study Chair — Mersin University, Department of Respiratory Diseases; Demet Polat Yulug, Dr., Principal Investigator — Mersin University, Department of Respiratory Diseases
Locations (1):
- Mersin University Faculty of Medicine, Department of Respiratory Diseases, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crisafulli E, Pisi R, Aiello M, Vigna M, Tzani P, Torres A, Bertorelli G, Chetta A. Prevalence of Small-Airway Dysfunction among COPD Patients with Different GOLD Stages and Its Role in the Impact of Disease. Respiration. 2017;93(1):32-41. doi: 10.1159/000452479. Epub 2016 Nov 17. PMID 27852080
- [Background] Bonini M, Usmani OS. The role of the small airways in the pathophysiology of asthma and chronic obstructive pulmonary disease. Ther Adv Respir Dis. 2015 Dec;9(6):281-93. doi: 10.1177/1753465815588064. Epub 2015 Jun 2. PMID 26037949